CLINICAL TRIAL: NCT03534791
Title: Interventions for Increasing Volunteer Engagement in Knowledge Translation Activity of Translating Cochrane Plain Language Summaries: a Randomized Controlled Trial
Brief Title: Brief Reminders as Intervention for Greater Engagement of Cochrane Translators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Split, School of Medicine (Other)
Collaborators: Croatian Science Foundation (Other Government)
Responsible Party: Principal Investigator, Dalibora Behmen, Professor, University of Split, School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014- 09-7672
Record Dates: First submitted 2018-05-09; First posted 2018-05-23 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Knowledge Translation

STUDY DESIGN:
Intervention Model Description: All study participants who accept participation in the study will be initially assigned 3 PLSs, and subsequently they will be assigned more PLSs when they translated the previous ones. Intervention group will receive one customized e-mail reminder two weeks after the PLS assignment if they do not translate it within two weeks.
  Control group will receive no intervention, i.e. standard procedure. Participants in the control group will receive PLSs for translation, in the frequency they indicated, and they will not receive any reminders. They will be assigned new PLSs once they translate the ones that were previously assigned.
Who Masked: Participant, Outcomes Assessor
Masking Description: Study participants will be blinded to allocation. The author who will communicate with the participants will not be blinded. Other authors and outcome assessors who will analyze data will be blinded to allocation of study participants; anonymized data will be analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reminders (Experimental): Reminders customized for each PLS, containing a name of the PLS indicated in the message. If the participants do not translate PLS within 2 months from PLS assignment, we will stop sending them reminders and we will consider them as dropouts.
  Interventions: Other: Reminders
- Control group (No Intervention): Control group will receive no intervention, i.e. standard procedure. Participants in the control group will receive PLSs for translation, in the frequency they indicated, and they will not receive any reminders. They will be assigned new PLSs once they translate the ones that were previously assigned.

INTERVENTIONS:
Other: Reminders — Personalized email which will aim for reminding of the translator about the PLSs on hold.
  Arms: Reminders

SUMMARY:
The intervention will consist of reminders which will be send to the participants randomly via email, with aim to increase the frequency and amount of translated plain language summaries (PLS).

DETAILED DESCRIPTION:
All study participants who accept participation in the study will be initially assigned 3 PLSs, and subsequently they will be assigned more PLSs when they translated the previous ones. Intervention group will receive one customized e-mail reminder two weeks after the PLS assignment if they do not translate it within two weeks. If they still do not translate the PLS, they will receive another customized e-mail reminder after every two weeks until they translate the PLS or until we reach maximum of 4 bi-weekly reminders (at 2 weeks, 4 weeks, 6 weeks and 8 weeks post-assignment) or until participants indicate that they are unable to translate it anymore. Text of the reminder that will be sent to the study participants is available in Supplementary file 1. The reminders will be customized for each PLS, and they will contain a name of the PLS indicated in the message. If the participants do not translate PLS within 2 months from PLS assignment, we will stop sending them reminders and we will consider them as dropouts.

Control group will receive no intervention, i.e. standard procedure. Participants in the control group will receive PLSs for translation, in the frequency they indicated, and they will not receive any reminders. They will be assigned new PLSs once they translate the ones that were previously assigned.

All PLSs will be translated in Memsource, a translation management tool that Cochrane plans to start using since March 2018 for managing translation of summaries. Participants will be followed 6 months from the moment of allocation.

ELIGIBILITY:
Inclusion Criteria:

* adults ≥18 years who volunteered to translate Cochrane PLSs within the Croatian translation project.

Exclusion Criteria:

* none

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Number of translated PLSs within the 6 month follow-up | 6 months
  The number of translated PLSs will be scored in the six months period for a participant

SECONDARY OUTCOMES:
Number of translated PLSs after 3 months of follow up | 3 months
  The number of translated PLSs will be scored in the three months period for a participant
Time to submitting translation | 6 months
  The investigators will note the time needed to submit translation
Satisfaction with participation in the translation project | 6 months
  Likert type scale from 1 to 10 (ranging from 1-completely unsatisfactory to 10-completely satisfactory)
Loss of participants | 6 months
  Loss of participants from the trial at final follow-up of 6 months, defined as participants' message that they wish to stop translating during the trial period, without later messages during the trial that they wish to engage in translation again.

CONTACTS AND LOCATIONS:
Overall Officials: Dalibora Behmen, Professor, Principal Investigator — Researcher and administrator
Locations (1):
- University of Split School of Medicine, Split, Split-Dalmatia County, Croatia

IPD SHARING:
Plan to Share IPD: Yes
Raw data will be posted to the Figshare repository (https://figshare.com/)
Time Frame: Within 12 months from study completion. The data will remain in the public repository indefinitely.
Access Criteria: Open access, publicly available

REFERENCES:
- [Derived] Jakus D, Behmen D, Buljan I, Marusic A, Puljak L. Efficacy of reminders for increasing volunteer engagement in translating Cochrane plain language summaries: a pilot randomised controlled trial. BMJ Evid Based Med. 2021 Apr;26(2):49-50. doi: 10.1136/bmjebm-2020-111378. Epub 2020 Jul 7. PMID 32636205